CLINICAL TRIAL: NCT02340715
Title: Investigation on the Utility of Advanced MRI Imaging Methods for Radiation Therapy Treatment Planning
Brief Title: Advanced MRI Sequences for Radiation Therapy Treatment Planning
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, AhunbayE, Chief of Physics, Medical College of Wisconsin
Other Study IDs: Advanced MRI
Record Dates: First submitted 2014-09-10; First posted 2015-01-19 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Cancer
Keywords: Anal canal; Brain; Breast; Cervix; Esophagus; Gynecology; Head and Neck; Lung; Pancreas; Primary liver or liver metastases; Prostate cancer; Sarcoma
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI for treatment planning or follow up: MRI for treatment planning for radiation therapy or those who have completed treatment and are receiving follow up care.

SUMMARY:
The purpose of this study is to determine if it would be helpful to use advanced MRI imaging techniques to take additional views of the tumor target for radiation treatment planning or treatment follow-up MRI.

DETAILED DESCRIPTION:
The results of this research project will be used to establish a standard MRI protocol specific to each tumor or disease site. An MRI protocol is a list of MR image types that are acquired for each disease site. These images are used to generate the patient's treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years older of any race or gender with anal canal, brain, breast, cervix, esophagus, gynecology, head and neck, lung, pancreas, primary liver or liver metastases, prostate cancer or sarcoma either undergoing MRI scan for radiation treatment planning or a post treatment MRI
* Voluntarily signs an IRB approved consent form

Exclusion Criteria:

* Inability to obtain informed consent from the patient or their medical power of attorney
* Patients who are not undergoing MR for radiation treatment planning
* Patients who will not have MRI scans after treatment
* Patients with pacemakers or other non-MRI compatible metallic implants
* Pregnant women, by self report using a standard MRI questionnaire
* Patients who will not receive contrast agent as part of their standard MR, will participate only in the non-contrast portion of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are planning to have radiation therapy for their cancer.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Ahunbay, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khoo VS, Dearnaley DP, Finnigan DJ, Padhani A, Tanner SF, Leach MO. Magnetic resonance imaging (MRI): considerations and applications in radiotherapy treatment planning. Radiother Oncol. 1997 Jan;42(1):1-15. doi: 10.1016/s0167-8140(96)01866-x. PMID 9132820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 420 was the initial estimate but 158 subjects was the accrual
Pre-assignment Details: 158 subjects were enrolled.
Period: Overall Study
Arm/Group | MRI for Treatment Planning or Follow up
Started | 158 (158)
Completed | 158 (158)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MRI for Treatment Planning or Follow up
Number analyzed (Participants) | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants] — Enrollment open to both genders.
  Participants
    Female | 85
    Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Contributing MRI Data
Description: We tested these Advanced MR protocols to evaluate which ones would best visualize the target region. This helped us determine the optimum MR SIM protocols for different sites that became clinical standard.
Time Frame: up to 4 weeks from imaging
Measure: Count of Participants; unit: Participants
Groups:
- MRI for Treatment Planning or Follow up: Patients aged 18 years and older of any race or gender with brain, head and neck, breast, lung, cervix, sarcoma, pancreatic, or prostate cancer undergoing MRI scans for radiation treatment planning and/or treatment follow-up at FMLH.
Arm/Group | MRI for Treatment Planning or Follow up
Number analyzed (Participants) | 158
Participants | 158

ADVERSE EVENTS:
Arm/Group | MRI for Treatment Planning or Follow up
Serious Adverse Events (participants affected / at risk) | 0/158
Other Adverse Events (participants affected / at risk) | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes